CLINICAL TRIAL: NCT00260156
Title: A Clinical Study to Assess the Effect of Vildagliptin on Beta Cell Function in Drug Naive Patients With Type 2 Diabetes
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CLAF237A2381
Record Dates: First submitted 2005-11-29; First posted 2005-12-01 (Estimated); Last update posted 2020-12-17 (Actual); Status verified 2013-01

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: Type 2 diabetes; vildagliptin
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Vildagliptin

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- vildagliptin (Experimental)
  Interventions: Drug: vildagliptin
- Placebo (Placebo Comparator)
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: vildagliptin
  Arms: vildagliptin
Drug: placebo
  Arms: Placebo

SUMMARY:
This study is not being conducted in the United States. The purpose of this study is to assess the effect of vildagliptin, an unapproved drug, on various measures of pancreatic islet function in people with type 2 diabetes who have not previously been treated with drug therapy to lower their blood sugar.

ELIGIBILITY:
Inclusion Criteria:

* Not currently on drug therapy for type 2 diabetes
* Blood glucose criteria must be met

Exclusion Criteria:

* History of type 1 diabetes
* Evidence of significant diabetic complications
* Serious cardiovascular events within the past 6 months
* Other protocol-defined exclusion criteria may apply

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2005-11; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
Change from baseline in hyperglycemia and arginine-stimulated first phase insulin secretion at 52 weeks | 52 weeks

SECONDARY OUTCOMES:
Change from baseline in disposition index at 52 weeks | 52 weeks
Change from baseline in hyperglycemia and arginine stimulated second phase insulin secretion at 52 weeks | 52 weeks
Change in hyperglycemia-stimulated first phase insulin secretion at 52 weeks | 52 weeks
Change in hyperglycemia-stimulated second phase insulin secretion at 52 weeks | 52 weeks
Beta-cell function parameter derived from standard meal challenge | 52 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (1):
- Novartis Pharmaceuticals, Basel, Switzerland

REFERENCES:
- [Derived] Foley JE, Bunck MC, Moller-Goede DL, Poelma M, Nijpels G, Eekhoff EM, Schweizer A, Heine RJ, Diamant M. Beta cell function following 1 year vildagliptin or placebo treatment and after 12 week washout in drug-naive patients with type 2 diabetes and mild hyperglycaemia: a randomised controlled trial. Diabetologia. 2011 Aug;54(8):1985-91. doi: 10.1007/s00125-011-2167-8. Epub 2011 May 6. PMID 21547496
- See also: Results for CLAF237A2381 on the Novartis clinical trials website — https://www.novctrd.com/ctrdweb/trialresult/trialresults/pdf?trialResultId=2798